CLINICAL TRIAL: NCT03289923
Title: Concurrent fMRI-guided rTMS and Cognitive Therapy for the Treatment of Major Depressive Episodes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 170147; 17-M-0147
Record Dates: First submitted 2017-09-20; First posted 2017-09-21 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Major Depressive Disorder
Keywords: Transcranial Magnetic Stimulation (TMS); Major Depressive Disorder; Cognitive Therapy
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active TMS+ Cognitive Therapy (Experimental): active
  Interventions: Device: Active TMS + Cognitive therapy
- Sham TMS + Cognitive Therapy (Sham Comparator): inactive
  Interventions: Device: Sham TMS + Cognitive therapy

INTERVENTIONS:
Device: Sham TMS + Cognitive therapy — Placebo Transcranial Magnetic Stimulation with cognitive therapy
  Arms: Sham TMS + Cognitive Therapy
Device: Active TMS + Cognitive therapy — Active Transcranial Magnetic Stimulation with cognitive therapy.
  Arms: Active TMS+ Cognitive Therapy

SUMMARY:
Background:

Repetitive transcranial magnetic stimulation (rTMS) is a treatment for depression. It stimulates the brain. Researchers want to see if using magnetic resonance imaging (MRI) scans helps locate the best area for rTMS in each person. They also want to find other ways to make it more effective.

Objective:

To study the effects of combining MRI- guided transcranial magnetic stimulation (TMS) and talk therapy on the brain in people with depression.

Eligibility:

Adults ages 18-75 with a major depressive disorder and current depression. If taking an antidepressant, should have been doing so for at least 4 weeks.

Design:

Participants will be screened with medical and psychiatric history, psychiatric evaluation, physical exam, and blood and urine tests.

Phase 1 is 1-4 visits in 1 week. Participants will have:

* Brain MRI. Participants will lie on a table in a scanner.
* Questions about their medical history and psychology symptoms
* Tests of mood and thinking
* Tests of brain activity. Participants may do tasks during these tests:

  * A cone with magnetic detectors is put on the head.
  * A cap with electrodes is put on the scalp.
  * TMS. A brief electrical current passes through a wire coil on the scalp.
  * A metal disk will be placed on the arm. A nerve will be stimulated with a small electrical shock.

Phase 2 is about 6 to 7 weeks.

* There will be 30 daily sessions of combined therapy and repetitive TMS (rTMS) for 6 weeks.
* Participants will receive rTMS and another therapy by computer.
* For rTMS, repeated pulses will pass through the coil.
* This is followed by up to 3 additional visits, when:

  * Participants will repeat Phase 1 tests
* Participants will rate their depression symptoms.

Phase 3 is 3 visits over 3 months. Participants will rate their depression symptoms and repeat some of the previous questionnaires and tests of mood and thinking.

DETAILED DESCRIPTION:
Objective

Despite the growing use of repetitive transcranial magnetic stimulation (rTMS) as a treatment for unipolar major depression, its typical effect sizes have been modest, and both methodological and conceptual challenges remain regarding how to optimize its efficacy. Two key elements have been missing from current work: first, to take an RDoC approach and link the treatment to a comprehensive model of the neurocircuitry underlying depression, where applying such a model to personalize the site of stimulation is likely to significantly improve the efficacy of rTMS; and second, to maximize neural changes to the engaged depression network by utilizing cognitive paired associate stimulation (C-PAS), a technique we have developed over the last decade in which noninvasive stimulation is applied to the targeted region while the circuit is engaged in processing related to desired behavior (here, through the simultaneous use of cognitive behavioral therapy). The concurrent firing in the emotional regulation circuit caused by TMS pulses and by the CBT will lead to neural plasticity according to the Hebbian conception of fire together, wire together, while repeated stimulation over the course of multiple TMS sessions will induce neuroplasticity to accelerate and strengthen those changes, which are expected to be therapeutic. We thus intend to test a novel integrative multimodal treatment for MDD consisting of a theory-based protocol for individualized optimization of rTMS site of stimulation plus concurrent behavioral interventions targeting the same dysfunctional neural circuitry. Our targeting procedure is based on recent developments in the psychology and neurobiology of self-regulation which offer a promising conceptual framework for identifying neural network mechanisms of action in rTMS for depression, as well as for developing guidelines for individualized rTMS treatment. As preliminary data, we report initial feasibility data from a clinical paradigm in which five adults with major depressionreceived TMS to the left middle frontal gyrus targeted on an individual basis using fMRI, while simultaneously receiving a previously validated self-regulation-based psychotherapy. Here, we will test this individualized method in a larger randomized trial.

Study Population

The study population will consist of 50 individuals between the 18 and 65 years of age, with a diagnosis of treatment-resistant Major Depressive Disorder (MDD).

Study Design

This single site study is a proof-of-concept clinical trial to test both functional states associated with an antidepressant response to a six week course of C-PAS using concomitant SST and 10 Hz rTMS neuronavigated to left DLPFC, as well as the feasibility and safety of such a course for long-term improvement in depressive symptoms. The proposed study will be conducted over 3 phases. Phase I will consist of screening, consent, and baseline measures. Screening will occur under the ETPB screening protocol (01-M-0254). Phase II will consist of a 6-week double-blind sham controlled trial of neuronavigated TMS cognitive therapy. Participants will be randomized to two groups, receiving either Active or Sham fMRI-guided-TMS, while involved in a cognitive therapy session. Subjects will participate in 30 daily sessions over 6 weeks, with MRI sessions both prior to and immediately after the course of TMS. Additionally, MEG may optionally be performed at baseline, immediately after the first TMS/SST session, and immediately after the entire course of TMS, and an optional battery of TMS/EEG excitability and plasticity measures may be performed pre- and post-TMS/SST course. In Phase III, the study team will provide standard of care for depression for up to three months, and will prescribe a relapse prevention strategy, in consultation with the referring physician, including TMS (which is consistent with standard of care).

Outcome Measures

Primary outcome measures are change in magnitude of BOLD signal recorded in pre- and post-TMS course MRI sessions, in the DLPFC region targeted with TMS based on individual activations in that region found at baseline using the priming task, and pre- and post-TMS course connectivity changes between DLPFC (measured with DTI and resting state functional connectivity), and other regions associated with the emotional regulation network, specifically OFC, medial PFC, precuneus, and ACC. Pre and post TMS course change in depression severity scores (HDRS, MADRS) will also be found, in order to look for correlations with these MRI measures. Secondary outcome measures will be ratings from the BSL, C-SSRS, CTQ, HAM-A, NIH-BFI, PANAS, RBANS, RRS, SHAPS, and TLEQ, as well as electrophysiological changes using MEG and EEG measures.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. 18 to 75 years of age.
  2. Use of effective method of birth control for women able to become pregnant
  3. English speaker
  4. Major Depressive Episode Diagnosis, and Severity:

     1. Subjects will meet the DSM-IV-TR primary diagnosis of initial or recurrent Major Depressive Disorder by DSM-IV-TR criteria
     2. HAM-D score > 17 and Item 1 score greater than or equal to 2. Alternatively: At the initial screening and beginning of Phase II, subjects must have a baseline score on the MADRS >= 20 and YMRS of < 12.
  5. Current or past history of lack of response to at least one adequate antidepressant trial, operationally defined using the Antidepressant Treatment History Form (ATHF); a failed adequate trial of ECT would count as an adequate antidepressant trial (unless the ECT occurred within the last year, in which case the participant will be excluded).
  6. If currently on a stable dose of antidepressant medication, the dosage has been unchanged for at least four weeks prior to study entry. The medication must be continued, and at the same dosage throughout study participation.
  7. Each subject must have a level of understanding sufficient to agree to all required tests and examinations and sign an informed consent document.
  8. All subjects must have undergone a screening assessment under protocol 01-M-0254, The Evaluation of Patients with Mood and Anxiety Disorders and Healthy Volunteers .
  9. Subjects are willing and able to adhere to the intensive treatment schedule and all required study visits.

EXCLUSION CRITERIA:

1. Pregnant or nursing women or women who plan to become pregnant in the next 20 weeks while in the study.

   Persons who are able to get pregnant must be willing to use at least one form of effective birth control during the entire period of study participation (or until last clinical labs and rating) and have a negative pregnancy test at screening.
2. Current or recent (within the past 6 months) diagnosis of substance abuse or dependence (excluding nicotine and caffeine)
3. Past or current history of tinnitus
4. Non English speaker
5. Unable to understand or complete study tasks and instructions
6. History of seizure except those therapeutically induced by ECT (childhood febrile seizures are acceptable and these subjects may be included in the study), history of epilepsy in self or first degree relatives, stroke, brain surgery, participants with history of any head trauma within 6 months of screening, or beyond 6 months prior to screening, history of head trauma with evidence of traumatic abnormality appearing on their brain scan, or with loss of consciousness >5 min, or with other sequelae, excluding headache, lasting > 24 hours will not be included in the study.
7. Diagnosed with the following conditions (current unless otherwise stated):

   1. Any other current primary Axis I mood or psychotic disorder, including bipolar disorder, with the exception of most anxiety disorders (including generalized anxiety disorder (GAD), social anxiety disorder (also known as social phobia), specific phobia, panic disorder with and without agoraphobia, posttraumatic stress disorder (PTSD), anxiety secondary to medical condition, acute stress disorder (ASD)), although with obsessive-compulsive disorder (OCD) and substance-induced anxiety disorder excluded. While these anxiety disorders can be comorbid, they must be stable and the MDD must be the primary diagnosis.
   2. Depression secondary to a general medical condition, or substance-induced.
   3. Any bipolar disorder or psychotic disorder (lifetime), including schizoaffective disorder, or major depression with psychotic features in this or previous episodes.
   4. Eating disorder (current or within the past year).
   5. Obsessive compulsive disorder (lifetime).
   6. Subjects meeting criteria for Axis II cluster A or B diagnosis based upon DSM-IV TR criteria, which in the judgment of the Investigator may hinder the subjects in completing the procedures required by the study protocol.
8. Subjects currently engaged or planning to engage in other treatment during the course of Phases I and II of the study (including behavior therapy, or other types of individual, family, or group psychotherapy/counseling), or subjects planning to start an antidepressant medication during the course of Phases I and II.
9. Increased risk of seizure for any reason, including prior diagnosis of increased intracranial pressure (such as after large infarctions or trauma), or currently taking medication that, in the opinion of the investigator, significantly lowers the seizure threshold.
10. Subjects with an unstable or serious medical or neurological disorder.
11. Presence of any medical illness likely to alter brain morphology and/or physiology (e.g., hypertension, diabetes) unless if controlled by medications.
12. Presence of any implants, prosthesis, or other permanent alteration of the body that, in the opinion of the investigator, would be unsafe with MRI or TMS or that would produce an artifact that would compromise the integrity of data.
13. Subjects who have hearing loss that has been clinically evaluated and diagnosed
14. Participants who are uncomfortable in small closed spaces (have claustrophobia), unable to lie comfortably supine for up to 90 minutes, and would feel uncomfortable in the MRI machine (for subjects doing imaging component of the study only).
15. Subjects with any of the following treatment histories:

    1. Lifetime history of TMS treatment.
    2. Lifetime history of treatment with Deep Brain Stimulation or Vagus Nerve Stimulation.
    3. Use of any investigational drug or device within 4 weeks of starting the study.
16. Clinically significant abnormal lab tests
17. Positive HIV test
18. Subjects who, in the investigator s judgment, pose a current serious suicidal or homicidal risk.
19. A current NIMH employee/staff or their immediate family member.
20. A positive test for COVID-19 or symptoms consistent with COVID-19 infection
21. Subjects who have allergies to lidocaine or previous adverse reaction to lidocaine.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2025-11-20 (Actual); Study Completion 2025-11-20 (Actual)

PRIMARY OUTCOMES:
Change in magnitude of Bold signal | 6 weeks after initiating intervention
  change in magnitude of BOLD signal with fMRI bold signal from DLPFC

SECONDARY OUTCOMES:
Electrophysiological changes using MEG and EEG measures | 6 weeks after initiating intervention
  Recordings of brain activity
Clinical Rating Scales: BSL, C-SSRS, CTQ, HAM-A, NIH-BFI, PANAS, RBANS, RRS, SHAPS, and TLEQ, | Variable: some 6 weeks after initiating intervention; others weekly
  Clinical symptom scales from which we derive scores

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Zarate, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-M-0147.html